CLINICAL TRIAL: NCT03350386
Title: Drug-drug Interaction Study to Evaluate the Pharmacokinetics and Safety of FYU-981 and Oxaprozin in Healthy Male Adults Subjects
Brief Title: Drug-drug Interaction Study of FYU-981 and Oxaprozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-017
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — dotinurad; Oxaprozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose (Experimental): Single administration of FYU-981
  Interventions: Drug: FYU-981
- Concomitant administration (Experimental): Concomitant administration of FYU-981 with oxaprozin at steady state
  Interventions: Drug: FYU-981; Drug: Oxaprozin

INTERVENTIONS:
Drug: FYU-981 — Single administration
Drug: Oxaprozin — Repeated administration
  Arms: Concomitant administration

SUMMARY:
This is an open-label, 2-period add-on study to assess the drug-drug interaction between FYU-981 and oxaprozin. The purpose of this study is to investigate the pharmacokinetics of each period in a single administration of FYU-981 and concomitant administration of FYU-981 with oxaprozin at steady -state in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy subjects
* Body mass index: >=18.5 and <25.0

Exclusion Criteria:

* Subject with any disease or any history of disease that might be unsuitable for participation in the clinical study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 48 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 48 hours
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 48 hours
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 48 hours
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (kel: Elimination rate constant) | 48 hours
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (MRT: Mean residence time) | 48 hours
Safety (Incidence of treatment-emergent adverse event) | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Nagasawa Katsuaki, Study Director — Clinical Research Department
Locations (1):
- P-One Clinic, Hachiōji, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furihata K, Nagasawa K, Hagino A, Kumagai Y. A drug-drug interaction study of a novel, selective urate reabsorption inhibitor dotinurad and the non-steroidal anti-inflammatory drug oxaprozin in healthy adult males. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):36-43. doi: 10.1007/s10157-020-01855-2. Epub 2020 Feb 19. PMID 32076889